CLINICAL TRIAL: NCT03100149
Title: A Randomized, Double-Blind, Placebo-Controlled, 52-Week Phase II Study to Evaluate the Efficacy of Intravenous RO7046015/Prasinezumab (PRX002) in Participants With Early Parkinson's Disease With a 11-Year All-Participants-on-Treatment Extension
Brief Title: A Study to Evaluate the Efficacy of Prasinezumab (RO7046015/PRX002) in Participants With Early Parkinson's Disease
Acronym: PASADENA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Prothena Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP39529; 2017-000087-15 (EudraCT Number); 2023-504472-24-00 (EU CTIS Number)
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: RO7046015 High Dose (Experimental): Participants will receive RO7046015 at high dose level as intravenous (IV) infusion every 4 weeks (Q4W) up to 52 weeks in Part 1.
  Interventions: Drug: RO7046015
- Part 1: RO7046015 Low Dose (Experimental): Participants will receive RO7046015 at low dose level as IV infusion Q4W up to 52 weeks in Part 1.
  Interventions: Drug: RO7046015
- Part 1: Placebo (Placebo Comparator): Participants will receive placebo as IV infusion Q4W up to 52 weeks in Part 1.
  Interventions: Drug: Placebo
- Part 2: RO7046015 High Dose (Experimental): Part 1 RO7046015 high dose group participants and placebo group participants randomized to high dose level will receive RO7046015 at high dose level as IV infusion Q4W for additional 52 weeks in Part 2.
  Interventions: Drug: RO7046015
- Part 2: RO7046015 Low Dose (Experimental): Part 1 RO7046015 low dose group participants and placebo group participants randomized to low dose level will receive RO7046015 at low dose level as IV infusion Q4W for additional 52 weeks in Part 2.
  Interventions: Drug: RO7046015
- Part 3: RO7046015 Low Dose (Experimental): All participants who complete Part 1 and Part 2 will receive monthly IV infusions of RO7046015.
  Interventions: Drug: RO7046015

INTERVENTIONS:
Drug: RO7046015 — RO7046015 will be administered at dose of 4500 milligrams (mg) for participants with body-weight greater than or equal to (>/=) 65 kilograms (kg) or 3500 mg for participants with body-weight less than (<) 65 kg.
  Other Names: PRX002; prasinezumab
  Arms: Part 1: RO7046015 High Dose; Part 2: RO7046015 High Dose
Drug: RO7046015 — RO7046015 will be administered at dose of 1500 mg to all participants in the indicated arm.
  Other Names: PRX002; prasinezumab
  Arms: Part 1: RO7046015 Low Dose; Part 2: RO7046015 Low Dose; Part 3: RO7046015 Low Dose
Drug: Placebo — RO7046015 placebo will be administered to all participants in the indicated arm.
  Arms: Part 1: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled, Phase 2 study will evaluate the efficacy of intravenous prasinezumab (RO7046015/PRX002) versus placebo over 52 weeks in participants with early Parkinson's Disease (PD) who are untreated or treated with monoamine oxidase B (MAO-B) inhibitors since baseline. The study will consist of three parts: a 52-week, double-blind, placebo-controlled treatment period (Part 1) after which eligible participants will continue into an all-participants-on-treatment blinded dose extension for an additional 52 weeks (Part 2). Participants who complete Part 2 (including the 12-week treatment-free follow up visit assessing long term safety and efficacy of RO7046015) will be offered participation in Part 3 open-label extension (all-participants-on-RO7046015-treatment) for an additional 520 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD with bradykinesia plus one of the other cardinal signs of PD (resting tremor, rigidity) being present, without any other known or suspected cause of PD untreated or treated with MAO-B inhibitor
* Body weight range between: >/=45 kg/ 99 pounds (lbs) and less than or equal to (</=) 110 kg/242 lbs
* Body mass index (BMI) of 18 to 34 kilograms per meter-squared (kg/m^2)
* A diagnosis of PD for 2 years or less at screening
* Hoehn and Yahr Stage I or II
* A screening brain DaT-SPECT consistent with PD (central reading)
* Clinical status does not require dopaminergic PD medication and is not expected to require dopaminergic treatment within 52 weeks from baseline
* If presently being treated for PD, a stable dose of MAO-B inhibitor (rasagiline or selegiline) for at least 90 days prior to baseline and not expected to change within 52 weeks
* For women of childbearing potential: use of highly effective contraceptive methods (that result in a failure rate of <1 percent [%] per year) during the treatment period and for at least 30 days (or longer if required by local regulations) after the last dose of study drug
* For men with female partners of childbearing potential or pregnant female partners, must use a condom during the treatment period and for at least 30 days (or longer if required by local regulations) after the last dose of study drug to avoid exposing the embryo. Men must refrain from donating sperm during this same period. The female partners should use a contraception method with a failure rate of <1% per year during the treatment period and for at least 30 days (or longer if required by local regulations) after the last dose of study drug. Use of contraceptive measures is not required for male participants enrolled in Part 3.

Exclusion Criteria:

* Medical history indicating a Parkinson syndrome other than idiopathic PD, including but not limited to, progressive supranuclear gaze palsy, multiple system atrophy, drug-induced parkinsonism, essential tremor, primary dystonia
* Known carriers of certain familial PD genes (as specified in study protocol)
* History of PD related freezing episodes or falls
* A diagnosis of a significant CNS disease other than Parkinson's disease; history of repeated head injury; history of epilepsy or seizure disorder other than febrile seizures as a child
* Mini Mental State Examination (MMSE) </=25
* Reside in a nursing home or assisted care facility
* History of or screening brain magnetic resonance imaging (MRI) scan indicative of clinically significant abnormality
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study or interfere with the participant's ability to comply with study procedures or abide by study restrictions, or with the ability to interpret safety data
* Any significant cardiovascular condition
* Any significant laboratory abnormality
* Lactating women
* Prior treatment with dopaminergic medication (for example, levodopa or a dopaminergic agonist) with no clinical treatment response or a clinical treatment response inconsistent with PD (for example, absence of observable response to a sufficiently high-dose of levodopa [i.e., ≥ 600 mg/day])
* Use of any of the following: catechol-O-methyl transferase (COMT) inhibitors (entacapone, tolcapone), amantadine or anticholinergics, or dopaminergic medication (levodopa and both ergot and non-ergot [pramipexole, ropinirole, rotigotine] dopamine agonists) for more than a total of 60 days or within 60 days of baseline
* Anti-epileptic medication for non-seizure-related treatment which has not remained stable for at least 60 days prior to baseline
* Anti-depressant or anxiolytic use that has not remained stable for at least 90 days prior to baseline. The use of fluoxetine and fluvoxamine is not permitted. For patients treated with a MAO-B inhibitor and an antidepressant (except fluoxetine and fluvoxamine), a 6-month period of stable and tolerated dosing before baseline is required.
* Use of any of the following within 90 days prior to baseline: antipsychotics (including clozapine and olanzapine), metoclopramide, alpha methyldopa, clozapine, olanzapine, flunarizine, amoxapine, amphetamine derivatives, reserpine, bupropion, buspirone, cocaine, mazindol, methamphetamine, methylphenidate, norephedrine, phentermine, phenylpropanolamine, and modafinil
* Participated in an investigational drug, device, surgical , or stem cell study in PD
* Any prior treatment with an investigational PD-related vaccine (including active immunization or passive immunotherapy with monoclonal antibodies).
* Prior participation in any RO7046015 or PRX002 study
* Receipt of any non-PD investigational product or device, or participation in a non-PD drug research study within a period of 30 days (or 5 half-lives of the drug, whichever is longer) before baseline
* Receipt of any monoclonal antibody or an investigational immunomodulator within 180 days (or 5 half-lives, whichever is longer) before baseline
* Immunomodulating drugs within 30 days prior to baseline
* Allergy to any of the components of RO7046015 such as citrate, trehalose and polysorbate (Tween) 20 or a known hypersensitivity or an Infusion-related reaction (IRR) to the administration of any other monoclonal antibody
* Any contraindications to obtaining a brain MRI. Patients with a hypersensitivity to iodine may receive an alternative thyroid blocking agent.
* For participants consenting to provide optional cerebrospinal fluid (CSF) samples by lumbar puncture (LP): LP will only be performed if the participant does not have any contraindication to undergoing an LP
* Donation of blood over 500 milliliters (mL) within three months prior to screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2031-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (26):
  - Uab Medicine, Birmingham, Alabama
  - Barrow Neurology Clinics, Phoenix, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - USC Keck Medical Center of USC, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Associated Neurologists of Southern CT PC, Fairfield, Connecticut
  - Molecular Neurolmaging, New Haven, Connecticut
  - Aventura Neurologic Associates, Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - USF Parkinsons Disease and Movement Disorders Center, Tampa, Florida
  - Northwestern University, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Corewell Health Neurology and Epilepsy - Beltline, Grand Rapids, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Oregon Health & Science Uni, Portland, Oregon
  - UNIVERSITY of PENNSYLVANIA, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Vermont Medical Center, Burlington, Vermont
- Medizinische Universität Innsbruck, Innsbruck, Austria
- France (11):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - Hôpital Michallon - Centre d'Investigation Clinique, Grenoble
  - hopital de la Timone, Marseille
  - CHU de Nice Hopital Pasteur, Nice
  - Hopital Pitie-Salpetriere APHP, Paris
  - CHU Poitiers, Poitiers
  - CHU Rouen Charles Nicolle, Rouen
  - CHU de Nantes - Hopital Laennec, Saint-Herblain
  - CIC - Hôpital Purpan, Toulouse
- Germany (8):
  - Klinik fur Neurologie, Berlin
  - Heinrich-Heine Universitätsklinik Düsseldorf, Düsseldorf
  - Paracelsus Elena Klinik Kassel, Kassel
  - Klinik und Poliklinik für Neurologie Universitätsklinikum, Leipzig
  - Philipps Universität Marburg, Marburg
  - DZNE Clinical Trial Unit, München
  - Universitaettsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Spain (9):
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Policlínica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Fundacion Hospital de Alcorcon, Alcorcón, Madrid
  - Clinica Universidad de Navarra, Pamplona/iruña, Navarre
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Taylor KI, Lipsmeier F, Scelsi MA, Volkova-Volkmar E, Rukina D, Popp W, Lambrecht S, Anzures-Cabrera J, Summers D, Abt M, Monnet A, Kilchenmann T, Schjodt-Eriksen J, Essioux L, Kustermann T, Zago W, Svoboda H, Nikolcheva T, Postuma RB, Pagano G, Lindemann M; PASADENA Investigators; Prasinezumab Study Group. Exploratory digital outcome measures of motor sign progression in Parkinson's disease patients treated with prasinezumab. NPJ Digit Med. 2025 Jun 16;8(1):365. doi: 10.1038/s41746-025-01572-8. PMID 40523921
- [Derived] Pagano G, Monnet A, Reyes A, Ribba B, Svoboda H, Kustermann T, Simuni T, Postuma RB, Pavese N, Stocchi F, Brockmann K, Smigorski K, Gerbaldo V, Fontoura P, Doody R, Kerchner GA, Brundin P, Marek K, Bonni A, Nikolcheva T; PASADENA Investigators; Prasinezumab Study Group. Sustained effect of prasinezumab on Parkinson's disease motor progression in the open-label extension of the PASADENA trial. Nat Med. 2024 Dec;30(12):3669-3675. doi: 10.1038/s41591-024-03270-6. Epub 2024 Oct 8. PMID 39379705
- [Derived] Pagano G, Taylor KI, Anzures-Cabrera J, Marchesi M, Simuni T, Marek K, Postuma RB, Pavese N, Stocchi F, Azulay JP, Mollenhauer B, Lopez-Manzanares L, Russell DS, Boyd JT, Nicholas AP, Luquin MR, Hauser RA, Gasser T, Poewe W, Ricci B, Boulay A, Vogt A, Boess FG, Dukart J, D'Urso G, Finch R, Zanigni S, Monnet A, Pross N, Hahn A, Svoboda H, Britschgi M, Lipsmeier F, Volkova-Volkmar E, Lindemann M, Dziadek S, Holiga S, Rukina D, Kustermann T, Kerchner GA, Fontoura P, Umbricht D, Doody R, Nikolcheva T, Bonni A; PASADENA Investigators; Prasinezumab Study Group. Trial of Prasinezumab in Early-Stage Parkinson's Disease. N Engl J Med. 2022 Aug 4;387(5):421-432. doi: 10.1056/NEJMoa2202867. PMID 35921451
- [Derived] Lipsmeier F, Taylor KI, Postuma RB, Volkova-Volkmar E, Kilchenmann T, Mollenhauer B, Bamdadian A, Popp WL, Cheng WY, Zhang YP, Wolf D, Schjodt-Eriksen J, Boulay A, Svoboda H, Zago W, Pagano G, Lindemann M. Reliability and validity of the Roche PD Mobile Application for remote monitoring of early Parkinson's disease. Sci Rep. 2022 Jul 15;12(1):12081. doi: 10.1038/s41598-022-15874-4. PMID 35840753
- [Derived] Pagano G, Boess FG, Taylor KI, Ricci B, Mollenhauer B, Poewe W, Boulay A, Anzures-Cabrera J, Vogt A, Marchesi M, Post A, Nikolcheva T, Kinney GG, Zago WM, Ness DK, Svoboda H, Britschgi M, Ostrowitzki S, Simuni T, Marek K, Koller M, Sevigny J, Doody R, Fontoura P, Umbricht D, Bonni A; PASADENA Investigators; Prasinezumab Study Group. A Phase II Study to Evaluate the Safety and Efficacy of Prasinezumab in Early Parkinson's Disease (PASADENA): Rationale, Design, and Baseline Data. Front Neurol. 2021 Oct 1;12:705407. doi: 10.3389/fneur.2021.705407. eCollection 2021. PMID 34659081
- [Derived] Jankovic J, Goodman I, Safirstein B, Marmon TK, Schenk DB, Koller M, Zago W, Ness DK, Griffith SG, Grundman M, Soto J, Ostrowitzki S, Boess FG, Martin-Facklam M, Quinn JF, Isaacson SH, Omidvar O, Ellenbogen A, Kinney GG. Safety and Tolerability of Multiple Ascending Doses of PRX002/RG7935, an Anti-alpha-Synuclein Monoclonal Antibody, in Patients With Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2018 Oct 1;75(10):1206-1214. doi: 10.1001/jamaneurol.2018.1487. PMID 29913017
- See also: Pasadenastudy.com provides information about the Roche clinical trial NCT03100149 and molecule being investigated in Parkinson's Disease — https://forpatients.roche.com/en/trials/neurodegenerative-disorder/pd/a-study-to-evaluate-the-efficacy-of-ro7046015-in-participants-wi.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 57 sites in 5 different countries. 1 site had only 1 screen failure and no active participants were enrolled there.
Pre-assignment Details: A total of 316 participants were randomized with a 1:1:1 allocation between the treatment groups (Placebo, Low-Dose prasinezumab and High-Dose prasinezumab)
Groups:
- Part 1: Placebo: Participants received placebo as intravenous (IV) infusion every four weeks (Q4W) up to 52 weeks in Part 1.
  Part 2 of the study occurs from Weeks 56 to 104. Participants initially randomized to placebo during Part 1 of the study will be rerandomized to one of the two active doses using a 1:1 allocation ratio. Part 2 is followed by 12 week termination follow-up safety visit and then by Part 3. Part 3 will last 260 weeks plus 12 weeks termination follow-up safety visit in which all participants will receive the low dose.
- Part 1: RO7046015 Low Dose: Participants received RO7046015 at a low dose level (1500 mg; for all body weights) as an IV infusion Q4W up to 52 weeks in Part 1.
  Part 2 of the study occurs from Weeks 56 to 104. Participants initially randomized to the low dose group will remain on their dose as assigned in Part 1. Part 2 is followed by 12 week termination follow-up safety visit and then by Part 3. Part 3 will last 260 weeks plus 12 weeks termination follow-up safety visit in which all participants will receive the low dose.
- Part 1: RO7046015 High Dose: Participants received RO7046015 at a high dose level (3500 mg for body weight <65 kilogram (kg) or 4500 mg for body weight >=65 kg) as an IV infusion Q4W up to 52 weeks in Part 1.
  Part 2 of the study occurs from Weeks 56 to 104. Participants initially randomized to the high dose group will remain on their dose as assigned in Part 1. Part 2 is followed by 12 week termination follow-up safety visit and then by Part 3. Part 3 will last 260 weeks plus 12 weeks termination follow-up safety visit in which all participants will receive the high dose.
Period: Overall Study
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Started | 105 | 105 | 106
Completed (Completed Part 1) | 105 | 101 | 104
Not Completed | 0 | 4 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Participant Moved out of Country | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population includes all participants randomized in the study who received any amount of study drug treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose | Total
Number analyzed (Participants) | 105 | 105 | 106 | 316
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (8.7) | 60.3 (8.8) | 59.4 (9.8) | 59.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 35 | 103
  Male | 71 | 71 | 71 | 213
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  Black or African American | 0 | 2 | 0 | 2
  White | 91 | 83 | 89 | 263
  Unknown | 13 | 20 | 17 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score (Sum of Parts I, II, and III) at Week 52
Description: The MDS-UPDRS is a multimodal scale consisting of four parts. Part I assessed non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contains 6 questions and are assessed by the examiner (Range 0-24). Part IB contains 7 questions on non-motor experiences of daily living which was completed by the participant (Range 0-28). Part II assessed motor experiences of daily living (Range 0-52). It contained 13 questions completed by the participant. Part III assessed the motor signs of Parkinson's Disease (PD) and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. The MDS-UPDRS Total Score equals the sum of Parts I,II, and III (Range: 0-236). A higher score indicated more severe symptoms of Parkinson's disease.
Time Frame: From baseline to Week 52
Population: The modified intent-to-treat (mITT) population includes all participants randomized in the study who received any amount of study drug treatment. Assessments of participants who started symptomatic therapy were included in the analysis up to the day before symptomatic treatment started.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 76 | 74 | 73
Units on a scale | 9.37 (1.221) | 7.35 (1.225) | 8.75 (1.234)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.2385, Mixed Models Analysis; Difference in Adjusted Means = -2.02, 80% CI 2-sided [-4.21 to 0.18], Standard Error of Mean 1.71
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.7169, Mixed Models Analysis; Difference in Adjusted Means = -0.62, 80% CI 2-sided [-2.82 to 1.58], Standard Error of Mean 1.71

2. Secondary Outcome: Change From Baseline in the MDS-UPDRS Part IA, Part IB, Part I Total, Part II Total, Part III Total and Part III Subscores
Description: The MDS-UPDRS is a multimodal scale consisting of four parts. Part I assessed non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contains 6 questions and are assessed by the examiner (Range 0-24). Part IB contains 7 questions on non-motor experiences of daily living which was completed by the participant (Range 0-28). Part II assessed motor experiences of daily living (Range 0-52). It contained 13 questions completed by the participant. Part III assessed the motor signs of Parkinson's Disease (PD) and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. There are 4 subscores in Part III: Bradykinesia, Rigidity, Resting tremors and Axial symptoms. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I,II, and III (Range:0-236). A higher score indicated more severe symptoms of Parkinson's disease.
Time Frame: From baseline to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 76 | 74 | 73
Units on a scale
  Part IA | -0.19 (0.119) | -0.27 (0.119) | -0.10 (0.121)
  Part IB | 0.94 (0.247) | 0.90 (0.248) | 0.96 (0.251)
  Part I total | 0.77 (0.295) | 0.59 (0.297) | 0.89 (0.300)
  Part II total | 2.75 (0.373) | 3.09 (0.375) | 2.69 (0.376)
  Part III total | 5.57 (0.897) | 3.69 (0.900) | 4.55 (0.911)
  Part III subscore - rigidity | 0.61 (0.263) | 0.70 (0.265) | 0.86 (0.268)
  Part III subscore - bradykinesia | 2.79 (0.556) | 1.72 (0.560) | 2.35 (0.565)
  Part III subscore - resting tremor | 1.20 (0.231) | 0.59 (0.233) | 0.79 (0.234)
  Part III subscore - axial symptoms | 0.19 (0.077) | 0.11 (0.078) | 0.18 (0.079)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part IA; Test type: Superiority; p = 0.6116, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.08, 80% CI 2-sided [-0.30 to 0.13], Standard Error of Mean 0.165
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part IA; Test type: Superiority; p = 0.6188, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.08, 80% CI 2-sided [-0.13 to 0.30], Standard Error of Mean 0.165
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part IB; Test type: Superiority; p = 0.9062, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.04, 80% CI 2-sided [-0.48 to 0.40], Standard Error of Mean 0.345
Statistical Analysis 4: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part IB; Test type: Superiority; p = 0.9621, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.02, 80% CI 2-sided [-0.43 to 0.46], Standard Error of Mean 0.347
Statistical Analysis 5: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part I Total; Test type: Superiority; p = 0.6510, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.19, 80% CI 2-sided [-0.71 to 0.34], Standard Error of Mean 0.411
Statistical Analysis 6: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part I Total; Test type: Superiority; p = 0.7709, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.12, 80% CI 2-sided [-0.41 to 0.65], Standard Error of Mean 0.413
Statistical Analysis 7: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part II Total; Test type: Superiority; p = 0.5177, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.34, 80% CI 2-sided [-0.33 to 1.01], Standard Error of Mean 0.523
Statistical Analysis 8: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part II Total; Test type: Superiority; p = 0.9095, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.06, 80% CI 2-sided [-0.73 to 0.61], Standard Error of Mean 0.523
Statistical Analysis 9: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part III Total; Test type: Superiority; p = 0.1354, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -1.88, 80% CI 2-sided [-3.49 to -0.27], Standard Error of Mean 1.255
Statistical Analysis 10: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part III Total; Test type: Superiority; p = 0.4217, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -1.02, 80% CI 2-sided [-2.64 to 0.61], Standard Error of Mean 1.262
Statistical Analysis 11: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part III Subscore: Rigidity; Test type: Superiority; p = 0.8053, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.09, 80% CI 2-sided [-0.38 to 0.56], Standard Error of Mean 0.369
Statistical Analysis 12: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part III Subscore: Rigidity; Test type: Superiority; p = 0.4970, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.25, 80% CI 2-sided [-0.22 to 0.73], Standard Error of Mean 0.370
Statistical Analysis 13: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part III Subscore: Bradykinesia; Test type: Superiority; p = 0.1703, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -1.07, 80% CI 2-sided [-2.07 to -0.07], Standard Error of Mean 0.779
Statistical Analysis 14: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part III Subscore: Bradykinesia; Test type: Superiority; p = 0.5729, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.44, 80% CI 2-sided [-1.45 to 0.56], Standard Error of Mean 0.782
Statistical Analysis 15: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part III Subscore: Resting Tremor; Test type: Superiority; p = 0.0628, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.61, 80% CI 2-sided [-1.02 to -0.19], Standard Error of Mean 0.324
Statistical Analysis 16: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part III Subscore: Resting Tremor; Test type: Superiority; p = 0.2125, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.41, 80% CI 2-sided [-0.82 to 0.01], Standard Error of Mean 0.325
Statistical Analysis 17: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; MDS-UPDRS Part III Subscore: Axial Symptoms; Test type: Superiority; p = 0.4577, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.08, 80% CI 2-sided [-0.22 to 0.06], Standard Error of Mean 0.108
Statistical Analysis 18: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; MDS-UPDRS Part III Subscore: Axial Symptoms; Test type: Superiority; p = 0.9182, Mixed Models Analysis — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.01, 80% CI 2-sided [-0.15 to 0.13], Standard Error of Mean 0.109

3. Secondary Outcome: Change From Baseline in Dopamine Transporter Imaging With Single Photon Emission Computed Tomography (DaT-SPECT) Striatal Binding Ratio (SBR) in the Putamen Ipsilateral to the Clinically Most Affected Side
Description: DaT-SPECT (dopamine transporter imaging with single photon emission computed tomography) is a dopamine transporter SPECT imaging that uses a radioactive agent called 123^I-ioflupane to quantify the density of the dopamine transporters in the striatum. Changes from baseline to week 52 in DaT-SPECT striatal binding ratios (SBRs; reference region: occipital cortex) in the putamen ipsilateral to the clinically most affected side were analyzed.
Time Frame: From baseline to Week 52
Population: The mITT population includes all participants randomized in the study who received any amount of study drug treatment and had no symptomatic PD treatment. The analysis included all assessments regardless of symptomatic treatment intake.
Measure: Least Squares Mean (Standard Error); unit: Striatal Binding Ratio (SBR)
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 102 | 100 | 104
Striatal Binding Ratio (SBR) | -0.08 (0.018) | -0.10 (0.018) | -0.11 (0.018)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.3582, ANCOVA — Nominal p-values are displayed for descriptive purposes only; LS Means Difference = -0.02, 80% CI 2-sided [-0.05 to 0.01], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.1955, ANCOVA — Nominal p-values are displayed for descriptive purposes only; LS Means Difference = -0.03, 80% CI 2-sided [-0.06 to 0.00], Standard Error of Mean 0.02

4. Secondary Outcome: Change From Baseline in Montreal Cognition Assessment (MoCA) Total Score
Description: The Montreal Cognitive Assessment (MoCA) is a rapid screening that was developed to be more sensitive to participants presenting with mild cognitive complaints. It briefly assesses short term and working memory, visuospatial abilities, executive function, attention, concentration, language and orientation. Scores on the MoCA test range from 0-30. Higher scores are associated with better cognitive function.
Time Frame: From baseline to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 104 | 100 | 103
Units on a scale | 0.07 (0.177) | 0.30 (0.181) | 0.51 (0.178)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.3611, ANCOVA — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.22, 80% CI 2-sided [-0.09 to 0.54], Standard Error of Mean 0.245
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.0727, ANCOVA — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = 0.44, 80% CI 2-sided [0.13 to 0.75], Standard Error of Mean 0.243

5. Secondary Outcome: Change From Baseline in Clinical Global Impression of Improvement (CGI-I) Score
Description: The CGI-I was intended as a measure of change in health status. CGI-I scores ranged from 1 (very much improved) through to 7 (very much worse). For the CGI-I, participants were divided into one of two groups, Responders or Progressors. Responders were scored on a scale of 1-4 which was rated as "no change", "minimally improved", "much improved" or "very much improved." Progressors were scored on a scale of 5-7 which was rated as "minimally worse", "much worse" or "very much worse." The percentage of participants rated by CGI-I Scale grouping at week 52 was analyzed using a logistic regression model.
Time Frame: From baseline to Week 52
Population: The mITT population includes all participants randomized in the study who received any amount of study drug treatment. Assessments of participants who started symptomatic therapy were included in the analysis up to the day before symptomatic treatment started.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 76 | 72 | 72
Percentage of participants
  Progressors | 56.6 | 50.0 | 48.6
  Responders | 43.4 | 50.0 | 51.4
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.4265, Regression, Logistic — Nominal p-values are displayed for descriptive purposes only; Odds Ratio (OR) = 0.77, 80% CI 2-sided [0.50 to 1.18]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.4063, Regression, Logistic — Nominal p-values are displayed for descriptive purposes only; Odds Ratio (OR) = 0.76, 80% CI 2-sided [0.49 to 1.16]

6. Secondary Outcome: Change From Baseline in Patient Global Impression of Change (PGIC) Score
Description: The PGIC was intended as a measure of change in health state from the participants perspective. PGIC scores ranged from 1 (very much improved) through to 7 (very much worse). For the PGIC, participants were divided into one of two groups, Responders or Progressors. Responders were scored on a scale of 1-4 which was rated as "no change", "minimally improved", "much improved" or "very much improved." Progressors were scored on a scale of 5-7 which was rated as "minimally worse", "much worse" or "very much worse." The percentage of participants rated by PGIC Scale grouping at week 52 was analyzed using a logistic regression model.
Time Frame: From baseline to Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 74 | 73 | 71
Percentage of participants
  Progressors | 58.1 | 50.7 | 53.5
  Responders | 41.9 | 49.3 | 46.5
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.3847, Regression, Logistic — Nominal p-values are displayed for descriptive purposes only; Odds Ratio (OR) = 0.75, 80% CI 2-sided [0.48 to 1.15]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.7055, Regression, Logistic — Nominal p-values are displayed for descriptive purposes only; Odds Ratio (OR) = 0.88, 80% CI 2-sided [0.57 to 1.36]

7. Secondary Outcome: Change From Baseline in Schwab and England Activity of Daily Living (SE-ADL) Score
Description: The SE-ADL is a single item scale assessing Activities of Daily Living on a scale ranging from 0% (bedridden) to 100% (completely independent), using 10% intervals.
Time Frame: From baseline to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 104 | 102 | 103
Units on a scale | -1.83 (0.644) | -2.56 (0.650) | -2.50 (0.647)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.4142, ANCOVA — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.73, 80% CI 2-sided [-1.87 to 0.41], Standard Error of Mean 0.888
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.4486, ANCOVA — Nominal p-values are displayed for descriptive purposes only; Difference in Adjusted Means = -0.67, 80% CI 2-sided [-1.81 to 0.47], Standard Error of Mean 0.885

8. Secondary Outcome: Time to Worsening in Motor or Non-Motor Symptoms
Description: This outcome measure is defined as the time to between first dose of study medication and the date when the particiapnt increases in MDS-UPDRS Part I (Range 0-52) of 3 or more points, or in MDS-UPDRS Part II (Range 0-52) of 3 or more points, whichever comes first. A higher score indicated more severe motor signs of Parkinson's disease.
Time Frame: From baseline to Week 52
Population: as for outcome 3
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 105 | 105 | 106
Days | 174.0 [168.0 to 225.0] | 169.0 [117.0 to 173.0] | 170.0 [168.0 to 222.0]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.3769, Regression, Cox — Nominal p-values are displayed for descriptive purposes only; Hazard Ratio (HR) = 1.15, 80% CI 2-sided [0.94 to 1.42]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.1658, Regression, Cox — Nominal p-values are displayed for descriptive purposes only; Hazard Ratio (HR) = 1.25, 80% CI 2-sided [1.02 to 1.53]

9. Secondary Outcome: Time to Start of Dopaminergic Parkinson's Disease Treatment
Description: This endpoint is defined as the time between first dose of study medication and the date when the participant starts dopaminergic treatment.
Time Frame: From baseline to Week 52
Population: as for outcome 3
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 105 | 105 | 106
Days | NA [NA to NA] — The median time to start of treatment" would be the timepoint when more than 50% of all participants started the treatment. At the end of Week 52, less than 50% of the participants started the treatment, thus the median time to start of treatment was not estimable. | NA [NA to NA] — The median time to start of treatment" would be the timepoint when more than 50% of all participants started the treatment. At the end of Week 52, less than 50% of the participants started the treatment, thus the median time to start of treatment was not estimable. | NA [NA to NA] — The median time to start of treatment" would be the timepoint when more than 50% of all participants started the treatment. At the end of Week 52, less than 50% of the participants started the treatment, thus the median time to start of treatment was not estimable.
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: RO7046015 Low Dose; Test type: Superiority; p = 0.9542, Regression, Cox — Nominal p-values are displayed for descriptive purposes only; Hazard Ratio (HR) = 1.01, 80% CI 2-sided [0.77 to 1.33]
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: RO7046015 High Dose; Test type: Superiority; p = 0.4567, Regression, Cox — Nominal p-values are displayed for descriptive purposes only; Hazard Ratio (HR) = 0.84, 80% CI 2-sided [0.63 to 1.13]

10. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was any AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From baseline to Week 52
Population: All randomized participants receiving any dose of the study drug were included in the safety analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
Number analyzed (Participants) | 105 | 105 | 106
Percentage of participants
  AEs | 82.9 | 93.3 | 91.5
  SAEs | 4.8 | 6.7 | 7.5

11. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) Against RO7046015
Description: Samples of the participant's blood was taken to evaluate anti-drug antibodies (ADA). The number of ADA positive participants, Treatment-induced and Treatment-enhanced was reported. Treatment-induced = participants with ADA negative or missing data at baseline but develop an ADA response following exposure to the study drug. Treatment-enhanced = participants with ADA positive at baseline and the titre of one or more post-baseline samples is at least >=4 fold increase greater than the baseline titre sample.
Time Frame: Baseline, Pre-dose (0 hours) on Weeks 4, 20, 36, 52, 56, 68, 80, and 104; at early termination (up to Week 104), and follow-up (12 weeks after last dose up to Week 116)
Reporting Status: Not Posted, anticipated posting 2027-04

12. Secondary Outcome: Systemic Clearance (CL) of RO7046015
Description: Clearance is a measure of the rate at which a drug is removed from the body.
Time Frame: Predose (0 hours) and end of infusion (infusion length=2 hours or less) on Baseline, Weeks 4, 20, 36, 52, 56, 68, 80, and 104; at Day 7, Day 14, early termination (up to Week 104), and follow-up (12 weeks after last dose up to Week 116)
Reporting Status: Not Posted, anticipated posting 2027-04

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of RO7046015
Description: Volume of distribution is defined as the theoretical volume which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 12
Reporting Status: Not Posted, anticipated posting 2027-04

14. Secondary Outcome: Area Under the Serum Concentration-Time Curve (AUC) of RO7046015 Over the Dosing Interval
Description: AUC is defined as the measure of RO7046015 plasma concentration over time.
Time Frame: Baseline over the duration of the study
Reporting Status: Not Posted, anticipated posting 2027-04

15. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of RO7046015 at Steady-state
Description: Cmax is the maximum observed plasma concentration of RO7046015.
Time Frame: Baseline over the duration of the study
Reporting Status: Not Posted, anticipated posting 2027-04

16. Secondary Outcome: Minimum Observed Serum Concentration (Ctrough) of RO7046015 at Steady-state
Description: Cmin is the minimum observed plasma concentration of RO7046015.
Time Frame: Baseline over the duration of the study
Reporting Status: Not Posted, anticipated posting 2027-04

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: AEs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0.
Arm/Group | Part 1: Placebo | Part 1: RO7046015 Low Dose | Part 1: RO7046015 High Dose
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105 | 0/106
Serious Adverse Events (participants affected / at risk) | 5/105 | 7/105 | 8/106
Other Adverse Events (participants affected / at risk) | 57/105 | 67/105 | 69/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=105) | Part 1: RO7046015 Low Dose (N=105) | Part 1: RO7046015 High Dose (N=106)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=105) | Part 1: RO7046015 Low Dose (N=105) | Part 1: RO7046015 High Dose (N=106)
Constipation (Gastrointestinal disorders) | 6 (6) | 8 (8) | 10 (10)
Nausea (Gastrointestinal disorders) | 9 (10) | 5 (6) | 9 (16)
Nasopharyngitis (Infections and infestations) | 15 (19) | 20 (25) | 13 (17)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 4 (4) | 9 (11)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 5 (9) | 10 (15)
Infusion related reaction (Injury, poisoning and procedural complications) | 17 (29) | 20 (40) | 35 (115)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 7 (8) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (8) | 11 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 5 (6)
Headache (Nervous system disorders) | 10 (12) | 10 (19) | 12 (15)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 7 (7)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3) | 8 (9)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03100149/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT03100149/SAP_000.pdf